CLINICAL TRIAL: NCT01613846
Title: Phase III Randomized Sequential Open-label Study to Evaluate the Efficacy and Safety of Sorafenib Followed by Pazopanib Versus Pazopanib Followed by Sorafenib in the Treatment of Advanced / Metastatic Renal Cell Carcinoma
Brief Title: Phase III Sequential Open-label Study to Evaluate the Efficacy and Safety of Sorafenib Followed by Pazopanib Versus Pazopanib Followed by Sorafenib in the Treatment of Advanced / Metastatic Renal Cell Carcinoma (SWITCH-II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16037 / AN 33/11; 2011-004396-36 (EudraCT Number); NCT02083094 (obsolete NCT alias)
Record Dates: First submitted 2012-05-04; First posted 2012-06-07 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

ARMS (2):
- Sorafenib followed by pazopanib (Experimental): Sorafenib 400 mg bid orally until progression or intolerable toxicity, followed by pazopanib 800 mg once daily orally until progression or intolerable toxicity.
  During first- and second-line, treatment visits are scheduled in weeks 0,2,4,8,12, and every 4 weeks thereafter, with tumor assessments and electrocardiogram after every second cycle (every 8 weeks).
  Interventions: Drug: Sorafenib+Pazopanib
- Pazopanib followed by Sorafenib (Experimental): Pazopanib 800 mg once daily orally until progression or intolerable toxicity, followed by Sorafenib 400 mg bid orally until progression or intolerable toxicity:
  During first- and second-line, treatment visits are scheduled in weeks, 0,2,4,8,12, and every 4 weeks thereafter, with tumor assessments and electrocardiogram after every second cycle (every 8 weeks).
  Interventions: Drug: Pazopanib+Sorafenib

INTERVENTIONS:
Drug: Sorafenib+Pazopanib — Sorafenib (first-line) followed by Pazopanib (second-line)
  Arms: Sorafenib followed by pazopanib
Drug: Pazopanib+Sorafenib — Pazopanib (first-line) followed by Sorafenib (second-line)
  Arms: Pazopanib followed by Sorafenib

SUMMARY:
Sorafenib and pazopanib are both effective and promising treatments for advanced Renal Cell Carcinoma (RCC). Both drugs are registered for this indication. No prospective comparative data in advanced RCC (or other indications) have been published. A search in the clinicaltrials.gov database did not reveal any planned or ongoing studies. As sequential therapy is now the standard of treatment for advanced RCC it is important to evaluate in clinical trials what the value of different sequential strategies is. This needs to be done every time new agents are introduced into the treatment armamentarium. As there are no data yet on the sequential use of sorafenib followed by pazopanib or vice versa, this sequence, however, will most certainly be used in daily practice, it is required to examine efficacy and safety of this sequential approach in a clinical trial in a randomized setting.

Therefore, the investigators have designed an open randomized study in patients not previously treated for advanced RCC. Suitable patients will be randomized (1:1) in 2 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic / advanced RCC (all histologies), who are not suitable for cytokine therapy and for whom study medication constitutes first-line treatment. For cytokine- unsuitability at least one of the following criteria must be fulfilled*:

   * Age 66 to 88 years
   * Non-clear cell histology RCC
   * Intermediate risk according to MSKCC score
   * ECOG ≥ 1 and> 1 organ metastasis + < 24 months between diagnosis and establishing indication for interleukin-2-therapy
   * ECOG ≥ 1 and "unable to carry on normal activity or do active work" (Karnofsky Index 70%)
   * Creatinine ≥ 1x ULN and < 2x ULN
   * Total bilirubin ≥ 1x ULN and < 1.5x ULN
   * Present autoimmune disease
   * Patients who might require steroids
   * Hypersensitivity against cytokines
   * Severe organic disease, not interfering with other in-/exclusion criteria of the Switch-2 study
   * Non-symptomatic brain metastases
   * Severe lung disease (e.g. PAH, COPD) with Pa O2 < 60 mmHg on rest
2. Age ≥ 18 and ≤ 85 years
3. Karnofsky Index ≥ 70% (see appendix 15.1)
4. MSKCC prognostic score (2004), low or intermediate (see appendix 15.2)
5. Life expectancy of at least 12 weeks
6. Subjects with at least one uni-dimensional (for RECIST 1.1) measurable lesion. Lesions must be measured by CT/MRI- scan
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of therapy:

   * hemoglobin > 9.0 g/dl
   * absolute neutrophil count (ANC) > 1,500 µl
   * Platelet count ≥ 100,000 / µl
   * total bilirubin < 1.5x the upper limit of normal (Note: Subjects with Gilbert' Syndrome are eligible if their total bilirubin is < 3.0 X ULN and direct bilirubin ≤ 35 %).
   * ALAT and ASAT < 2.5x upper limit of normal (Note: concomitant elevations in bilirubin ans ASAT/ALAT above 1.0x upper limit of normal are not permitted).
   * Alkaline phosphatase < 4x upper limit of normal
   * PT-INR/aPTT < 1.2x upper limit of normal (Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that their INR is stable and within the recommended range for the desired level of anticoagulation and no prior evidence of underlying abnormality in these parameters exists).
   * Serum creatinine < 2x upper limit of normal
8. Written Informed Consent

Exclusion Criteria:

1. History of cardiac disease: congestive heart failure > NYHA class 2 or with LVEF at baseline echocardiography < 50%, (echocardiography is optional); active CAD (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
2. Uncontrolled hypertension (defined as blood pressure ≥ 150 mmHg systolic and/or ≥ 90 mmHg diastolic on medication).
3. History of HIV infection or chronic hepatitis B or C
4. 4. Active clinically serious infections (> grade 2 NCI-CTC version 4.03)
5. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
6. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
7. Patients with evidence or history of bleeding diathesis
8. History of organ allograft
9. Major surgery within 4 weeks of start of study
10. Autologous bone marrow transplant or stem cell rescue within 4 months before study start.
11. Any significant condition that increases the risk for bleeding, including, but not limited to active peptic ulcer disease, inflammatory bowel disease, known intraluminal or endobronchial metastatic lesions and/or lesions infiltrating major pulmonary vessels with risk of bleeding, presence of non-healing wound or trauma within 4 weeks prior to first dose of investigational drug
12. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep vein thrombosis (DVT) within the past 6 months (Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible)
13. Corrected QT Interval (QTc) > 480 msecs
14. Untreated hypothyroidism
15. Patients undergoing renal dialysis
16. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry
17. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures (with a Pearl Index < 1) during the course of the trial and 3 months after the completion of trial
18. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
19. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
20. Patients unable to swallow oral medications
21. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
22. Known allergy to Votrient or Nexavar (i.e. to active substance or one of the constituents)
23. Prior exposure to study drugs.
24. Investigational drug therapy within 4 weeks of study entry.
25. Use of biologic response modifiers, such as G-CSF and other hematopoietic growth factors, within 3 weeks of study entry
26. Radiotherapy within 3 weeks of start of study drug and planned radiotherapy during the study
27. Concomitant medication: Any condition at the discretion of the investigator that precludes compliance with concomitant therapy restrictions described below.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
To evaluate if progression-free survival from randomization to progression or death during second-line therapy (Total PFS) of sorafenib followed by pazopanib is non-inferior compared to pazopanib followed by sorafenib. | 4 years

SECONDARY OUTCOMES:
Time from randomization to progression during second-line therapy (total TTP) | 1 year
Time to first-line treatment failure (progression, death, discontinuation due to toxicity) descriptively in each arm | 1 year
PFS in first-line and second-line treatment, descriptively | 4 years
Overall survival, descriptively (data cut-off same as for primary endpoint | 4 years
Disease Control Rate (DCR); Response rates in first-line and in second-line (CR, PR, SD according to RECIST criteria) | 4 years
Health-related Quality of Life (FACIT-F, FKSI-10) | 4 years
Biomarker programme | 4 years
  Circulating tumor cells, Single Nucleotide Polymorphisms, Serum Protein Signatures
Safety and tolerability | 4 years
  Monitoring of adverse events, summaries and listings of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen E. Gschwend, Prof., Principal Investigator — Klinikum rechts der Isar, TU München
Locations (72):
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - A. ö. Bezirkskrankenhaus Kufstein, Kufstein
  - AKH Linz GmbH, Linz
  - LKH Salzburg, Salzburg
- Germany (62):
  - Universitätsklinikum Aachen, Urologische Klinik, Aachen
  - Gesundheitszentrum St. Marien GmbH, Amberg
  - Praxis für Urologie, Berlin
  - Charite Campus Virchow Klinikum / Klein. Für Innere Med / Onkologie/Hämatologie, Berlin
  - Gemeinschaftspraxis Pott / Tirier / Hannig - Onkologie, Bottrop
  - Urologie im Schlosscarrée Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Bethanien Krankenhaus Chemnitz gGmbH, Chemnitz
  - Überörtliche Gemeinschaftspraxis, Cologne
  - Onkologische Gemeinschaftspraxis Dörfel/Göhler, Dresden
  - Universitätsklinikum Carl Gustav Carus der Technischen Universität Dresden, Dresden
  - Urologische Gemeinschaftspraxis, Duisburg
  - Krankenhaus Düren gGmbH, Düren
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Urologische Facharztpraxis, Eisleben Lutherstadt
  - Urologie Neandertal - Ortsübergreifende Gemeinschaftspraxis für Urologie, Erkrath
  - Waldkrankenhaus St. Marien, Erlangen
  - St.-Antonius-Hospital in Eschweiler / Klinik f. Hämatologie und Onkologie, Eschweiler
  - Hämato-onkologische Gemeinschaftspraxis, Essen
  - Onkozentrum Freiberg, Freiberg
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - MVZ Osthessen GmbH, Fulda
  - Gem.praxis Dres. J. Wilke, H. Wagner - Hämatol.u.intern.Onkol. am Klinikum Fürth, Fürth
  - Onkologische Schwerpunktpraxis, Goslar
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - St. Antonius-Hospital Gronau GmbH, Gronau
  - Onkologische Schwerpunktpraxis, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Heidelberg, Klinik für Urologie, Heidelberg
  - Urologie-Heinsberg, Heinsberg
  - Onkologische Praxis, Hildesheim
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Jena, Klinik für Urologie, Jena
  - Praxis für Urologie, Lauenburg
  - Onkologische Schwerpunktpraxis Leer - Emden, Leer
  - MVZ Mitte/ MVZ Delitzsch GmbH, Leipzig
  - Universitätsklinikum Magdeburg A.ö.R, Magdeburg
  - Universitätsklinik Mannheim, Mannheim
  - Philips-Universität-Marburg, Urologie und Kinderurologie, Marburg
  - Praxis Markkleeberg, Markkleeberg
  - Kliniken Maria Hilf, Mönchengladbach
  - PUR/R Praxisklinik Urologie Rhein Rhur, Mühlheim
  - Klinikum r. d. Isar, Klinik für Urologie, München
  - Universitätsklinikum Münster , Klinik für Urologie, Münster
  - Eps- early phase solutions GmbH, Pößneck
  - Caritas Krankenhaus St. Josef, Regensburg
  - Universitätsklinikum Rostock, Rostock
  - Zentrum für Urologie und Onkologie, Rostock
  - Diakoniekrankenhaus Rotenburg (Wümme) gGmbH, Rotenburg (Wümme)
  - Klinikum Sindelfingen-Böblingen, Sindelfingen
  - Marienhospital / Innere Med III Onko Hämato Palliativm, Stuttgart
  - Eberhard-Karls-Universität Tübingen, Tübingen
  - Universitätsklinik Ulm, Ulm
  - Universitätsklinikum Ulm, Ulm
  - Praxis für Hämatologie und internistische Onkologie, Velbert
  - Klinikum Nordoberpfalz AG, Weiden
  - Gesellsch. z. Förd. Von Wissenschaft u.Qualitätssicherung i.d.ambul.Onkologie, Wiesbaden
  - Praxisgemeinschaft für Onkologie und Urologie, Wilhelmshaven
  - Gemeinschaftspraxis für Urologie, Wuppertal
  - Universitätsklinikum Würzburg, Würzburg
- Netherlands (6):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Spaarne Ziekenhuis, Hoofddorp
  - HAGA, The Hague
  - TweeSteden Ziekenhuis, Tilburg
  - VieCuri Medical Center, Venlo

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Retz M, Bedke J, Bogemann M, Grimm MO, Zimmermann U, Muller L, Leiber C, Teber D, Wirth M, Bolenz C, van Alphen R, De Santis M, Beeker A, Lehmann J, Indorf M, Frank M, Bokemeyer C, Gschwend JE. SWITCH II: Phase III randomized, sequential, open-label study to evaluate the efficacy and safety of sorafenib-pazopanib versus pazopanib-sorafenib in the treatment of advanced or metastatic renal cell carcinoma (AUO AN 33/11). Eur J Cancer. 2019 Jan;107:37-45. doi: 10.1016/j.ejca.2018.11.001. Epub 2018 Dec 7. PMID 30529901